CLINICAL TRIAL: NCT02052050
Title: Effectiveness of Core Stability Exercises on Abdominal Deep Muscles in Colorectal Cancer Survivors
Brief Title: Core Stability Program in Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Manuel Arroyo Morales, PhD, MD, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEI2013-MP-18
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal-neoplasms,deep-muscles of the back,rehabilitation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Core Stability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- core stability (Experimental): Stabilized muscle program will consist of two months of individual physical training that it will be conducted 3 times/week for 90 min each. A correct progression to improve stabilization of deep abdominal muscles will be made.
  Interventions: Other: core stability
- control group (No Intervention): usual care

INTERVENTIONS:
Other: core stability
  Arms: core stability

SUMMARY:
The purpose of this study is to determine the effects of physical training program to improve deep stabilizer muscle in colorectal cancer survivors

DETAILED DESCRIPTION:
Background: Colorectal cancer is the third most common cancer when considering both genders. Musculoskeletal alterations have been described related to techniques used during surgery, that it produces an inhibition of deep abdominal muscles. These muscles are in charge of lumbopelvic stabilization muscle linked to reduced ability to maintain independence in daily activity life that could have affected their quality of life

Objective: The aim objective will be evaluated short and long-term effects of physical activity program for muscle stabilization.

Methods: 20 colorectal cancer survivors will be recruited from the Department of Oncology of Clínico San Cecilio Hospital. Patients will be randomized in physical activity program group and usual care group. Physical activity groups will receive an eight week program form improve the muscle stabilization.

Discussion: Researchers attempts to increase the fitness level and reduce musculoskeletal disorders in colorectal cancer survivors through a physical activity interventions focusing in muscle stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients under partial colorectal resection to treat colon cancer
* Diagnosis of I, II or IIIa stage of colorectal cancer
* Completion of adjuvant therapy (except for hormone therapy)
* Medical clearance of participation

Exclusion Criteria:

Participants will be excluded if they presents with cancer recurrence or if they will have undergone previous abdominal surgeries or will be diagnosed with concomitant conditions, such as previous lower-back pain or musculoskeletal conditions (e.g., osteoarthritis, fibromyalgia or chronic fatigue syndrome).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Abdominal isometric endurance | Baseline- 8 weeks
  Isometric endurance of trunk flexors will be used to determine endurance strength of abdominal muscles. Patients will be laid supine, maintaining hips and knees bent at 90 degrees, feet flat approximately 30 inches from the buttocks and arms extended with hands on knees without actually touching. Patients will be instructed to separate the trunk from the stretcher to the inferior angle of the scapula and maintain this position as long as possible. Time (in seconds) will be measured until a maximum of 90 seconds

SECONDARY OUTCOMES:
Fatigue | Baseline- 8 weeks
  The Piper Fatigue Scale will be used for it measure. It scale includes 22 items and four dimensions (behavioural/severity, affective meaning, sensory and cognitive mood)
Body composition: | Baseline- 8 weeks
  It will be obtained with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea)
Pain: | Baseline- 8 weeks
  The participants will be completed a visual analogue scale to assess the presence of lower-back and/or abdominal pain. The Brief Pain Inventory (BPI) will be used to assess the interference and the experience of pain.
Static balance | Baseline- 8 weeks
  The Flamingo Test
Flexibility | Baseline- 8 weeks
  The "chair sit and reach test"
Functional capacity | Baseline- 8 weeks
  The 6-min walk test with treadmill (H-P-COSMOS for graphics; Germany)
Fitness perceived | Baseline- 8 weeks
  The International Fitness Scale (IFIS)
Lower back muscle strength | Baseline- 8 weeks
  dynamometer (TKK 5002 Back-A; Takey, Tokyo, Japan)

OTHER OUTCOMES:
Quality of life | Baseline- 8 weeks
Pressure Pain Thresholds | Baseline- 8 weeks
Muscle structure | Baseline- 8 weeks
  An ultrasound device (MyLab™ 25, Esaote Medical Systems, Genova, Italy) and a 12 MHz linear probe will be used in this study. The depth of internal and external oblique and transversus abdominis, and depth and width of lumbar multifidus will be captured when the patient will be relaxed at the end of the expiration movement.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero Villanueva, PhD, Study Chair — Universidad de Granada
Locations (1):
- University of Granada. Faculty of Health Sciences, Granada, Granada, Spain

REFERENCES:
- [Background] Temple PC, Travis B, Sachs L, Strasser S, Choban P, Flancbaum L. Functioning and well-being of patients before and after elective surgical procedures. J Am Coll Surg. 1995 Jul;181(1):17-25. PMID 7599766
- [Background] Slattery ML. Physical activity and colorectal cancer. Sports Med. 2004;34(4):239-52. doi: 10.2165/00007256-200434040-00004. PMID 15049716
- [Background] Cantarero-Villanueva I, Fernandez-Lao C, Cuesta-Vargas AI, Del Moral-Avila R, Fernandez-de-Las-Penas C, Arroyo-Morales M. The effectiveness of a deep water aquatic exercise program in cancer-related fatigue in breast cancer survivors: a randomized controlled trial. Arch Phys Med Rehabil. 2013 Feb;94(2):221-30. doi: 10.1016/j.apmr.2012.09.008. Epub 2012 Sep 24. PMID 23017985
- [Background] Cantarero-Villanueva I, Fernandez-Lao C, Del Moral-Avila R, Fernandez-de-Las-Penas C, Feriche-Fernandez-Castanys MB, Arroyo-Morales M. Effectiveness of core stability exercises and recovery myofascial release massage on fatigue in breast cancer survivors: a randomized controlled clinical trial. Evid Based Complement Alternat Med. 2012;2012:620619. doi: 10.1155/2012/620619. Epub 2011 Jul 17. PMID 21792370
- [Background] Fernandez-Lao C, Cantarero-Villanueva I, Fernandez-de-Las-Penas C, del Moral-Avila R, Castro-Sanchez AM, Arroyo-Morales M. Effectiveness of a multidimensional physical therapy program on pain, pressure hypersensitivity, and trigger points in breast cancer survivors: a randomized controlled clinical trial. Clin J Pain. 2012 Feb;28(2):113-21. doi: 10.1097/AJP.0b013e318225dc02. PMID 21705873
- [Derived] Cantarero-Villanueva I, Sanchez-Jimenez A, Galiano-Castillo N, Diaz-Rodriguez L, Martin-Martin L, Arroyo-Morales M. Effectiveness of Lumbopelvic Exercise in Colon Cancer Survivors: A Randomized Controlled Clinical Trial. Med Sci Sports Exerc. 2016 Aug;48(8):1438-46. doi: 10.1249/MSS.0000000000000917. PMID 27015381